CLINICAL TRIAL: NCT04568408
Title: Validation of the Quality of Sleep Data for Xiaomi Domestic Wristbands
Status: Completed | Type: Observational
Sponsor: Universidade da Coruña (Other)
Collaborators: Center on Information and Communication Technologies (Other); IMQ San Rafael (Unknown)
Responsible Party: Principal Investigator, Javier Pereira, Proffesor PhD, Universidade da Coruña
Other Study IDs: 2020/318
Record Dates: First submitted 2020-09-16; First posted 2020-09-29 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Sleep Disorder
Keywords: Sleep; Polysomnography; Occupational Performance; Participatory Health; Internet of Things; Wearables
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sleep study participants: Adults presenting sleep difficulties or poor sleep quality that are performed a Polisomnography study in a Sleep Unit at hospital.
  Interventions: Device: Xiaomi MiBand 5

INTERVENTIONS:
Device: Xiaomi MiBand 5 — Comparison of sleep-monitoring device against polysomnography (PSG)

SUMMARY:
Introduction: Polysomnography (PSG) is currently the accepted Gold Standard for sleep studies as it measures multiple variables that lead to a clear diagnosis of any sleep disorder. However, it has some clear drawbacks as it can only be performed by qualified technicians, has a high cost and complexity and is very invasive. In the last years, Actigraphy has been used along with PSG for sleep studies. In this study, the investigators intend to assess the capability of the new Xiaomi Mi Band 5 to be used as a sleep self-assessment tool for patients.

Objective: Determine whether sleep stages recorded by the new Xiaomi Mi Band 5 can effectively replace PSG sleep stages classification in patients that undergo a sleep study.

Methods and analysis: the study will be carried out with patients in a hospital from A Coruña (Galicia, Spain) that are > 18 years old. Patients who are performed a polysomnography test will be given the wearables so the investigators can record sleep stages with both techniques in order to compare both recordings afterwards.

This is an observational, analytic and longitudinal study. In other words, in this study different variables from the population of interest will be observed and recorded without any direct intervention, so as to establish causality associations between these variables. It is considered as longitudinal since a six-months tracking of the variables will be performed, continually (and sometimes occasionally) recording and monitoring sleep quality (wearable wristbands).

The data obtained from PSG and Xiaomi Mi Band 5 will be preprocessed and explored before extracting the features of interest for the study. Then, Paired sample T-Test will be performed to compare the means among the different variables, Bland-Altman plots will be used to assess the concordance between both techniques and, finally, Epoch by Epoch analysis will be performed to compare the classification of the sleep stages carried out by both PSG and Xiaomi.

DETAILED DESCRIPTION:
Introduction: Sleep disorders are becoming a widespread health problem within the general population. Beyond the tiredness itself, these disorders have been found to be related to physical and mental issues like cardiovascular pathologies, obesity, depression and anxiety. This makes clear the necessity of achieving a quality rest to prevent potential chronic diseases. On this issue, Polysomnography (PSG) is currently the accepted Gold Standard for sleep studies as it measures multiple variables that lead to a clear diagnosis of any sleep disorder. However, it has some clear drawbacks as it can only be performed by qualified technicians, has a high cost and complexity and is very invasive. In the last years, several studies that focus on validating wearable devices as useful sleep trackers have emerged. In this study, the investigators intend to assess the capability of the new Xiaomi Mi Band 5 to be used as a tool for sleep self-assessment for patients. The interest in studying this smartband is due to its low price and acceptance among the population. If this device proves to be a good sleep tracker, it would allow the population to assess their own sleep and consider if they need to visit their medical practitioner, which would improve the prognosis of any underlying condition they may be developing derived from their restlessness.

Objective: Determine whether sleep stages recorded by the new Xiaomi Mi Band 5 can effectively replace PSG sleep stages classification in patients that undergo a sleep study. The following features will be calculated for both devices: total sleep time, sleep efficiency, sleep latency and wake after sleep onset. Sleep stages will also be recorded.

Methods and analysis: the study will be carried out with patients in a hospital from A Coruña (Galicia, Spain) that are > 18 years old. Patients who are performed a polysomnography test will be given the wearables so the investigators can record sleep stages with both techniques in order to compare both recordings afterwards.

This is an observational, analytic and longitudinal study. In other words, in this study different variables from the population of interest will be observed and recorded without any direct intervention, so as to establish causality associations between these variables. It is considered as longitudinal since a six-months tracking of the variables will be performed, continually (and sometimes occasionally) recording and monitoring sleep quality (wearable wristbands).

The data obtained from PSG and Xiaomi Mi Band 5 will be preprocessed and explored before extracting the features of interest for the study. Then, Paired sample T-Test will be performed to compare the means among the different variables, Bland-Altman plots will be used to assess the concordance between both techniques and, finally, Epoch by Epoch analysis will be performed to compare the classification of the sleep stages carried out by both PSG and Xiaomi.

ELIGIBILITY:
Inclusion Criteria:

* Attending to the Sleep Unit to be perfomed a Polysomnography study
* Declaring a chronological age that is equal or higher than 18 years old

Exclusion Criteria:

* Having significant health complications that hinder active participation in the study
* Suffering from skin hypersensitivity or an allergic reaction due to the materials the wristbands that will be used in the study as measuring instruments are made of

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with a self-perception of sleep problems or poor quality of their sleep
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Sleep recording Reliability | 6 Months
  Assessment of sleep measurement and sleep stages classification

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pereira, PhD, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wade AG. The societal costs of insomnia. Neuropsychiatr Dis Treat. 2010 Dec 20;7:1-18. doi: 10.2147/NDT.S15123. PMID 21326650
- [Background] Chen JH, Waite L, Kurina LM, Thisted RA, McClintock M, Lauderdale DS. Insomnia symptoms and actigraph-estimated sleep characteristics in a nationally representative sample of older adults. J Gerontol A Biol Sci Med Sci. 2015 Feb;70(2):185-92. doi: 10.1093/gerona/glu144. Epub 2014 Sep 8. PMID 25199910
- [Background] Koffel E, McCurry SM, Smith MT, Vitiello MV. Improving pain and sleep in middle-aged and older adults: the promise of behavioral sleep interventions. Pain. 2019 Mar;160(3):529-534. doi: 10.1097/j.pain.0000000000001423. No abstract available. PMID 30562269
- [Background] Kurina LM, Thisted RA, Chen JH, McClintock MK, Waite LJ, Lauderdale DS. Actigraphic sleep characteristics among older Americans. Sleep Health. 2015 Dec;1(4):285-292. doi: 10.1016/j.sleh.2015.09.004. PMID 28815195
- [Background] Chamorro N, Sellares J, Millan G, Cano E, Soler N, Embid C, Montserrat JM. An integrated model involving sleep units and primary care for the diagnosis of sleep apnoea. Eur Respir J. 2013 Oct;42(4):1151-4. doi: 10.1183/09031936.00192812. No abstract available. PMID 24081767
- [Background] Merilahti J, Korhonen I. Association between Continuous Wearable Activity Monitoring and Self-Reported Functioning in Assisted Living Facility and Nursing Home Residents. J Frailty Aging. 2016;5(4):225-232. doi: 10.14283/jfa.2016.102. PMID 27883169
- [Background] Shelgikar AV, Anderson PF, Stephens MR. Sleep Tracking, Wearable Technology, and Opportunities for Research and Clinical Care. Chest. 2016 Sep;150(3):732-43. doi: 10.1016/j.chest.2016.04.016. Epub 2016 Apr 29. PMID 27132701
- [Background] Griessenberger H, Heib DP, Kunz AB, Hoedlmoser K, Schabus M. Assessment of a wireless headband for automatic sleep scoring. Sleep Breath. 2013 May;17(2):747-52. doi: 10.1007/s11325-012-0757-4. Epub 2012 Sep 21. PMID 22996794
- [Background] Lee PH, Suen LK. The convergent validity of Actiwatch 2 and ActiGraph Link accelerometers in measuring total sleeping period, wake after sleep onset, and sleep efficiency in free-living condition. Sleep Breath. 2017 Mar;21(1):209-215. doi: 10.1007/s11325-016-1406-0. Epub 2016 Sep 10. PMID 27614441
- [Background] Smith MT, McCrae CS, Cheung J, Martin JL, Harrod CG, Heald JL, Carden KA. Use of Actigraphy for the Evaluation of Sleep Disorders and Circadian Rhythm Sleep-Wake Disorders: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2018 Jul 15;14(7):1231-1237. doi: 10.5664/jcsm.7230. PMID 29991437
- [Background] Xie J, Wen D, Liang L, Jia Y, Gao L, Lei J. Evaluating the Validity of Current Mainstream Wearable Devices in Fitness Tracking Under Various Physical Activities: Comparative Study. JMIR Mhealth Uhealth. 2018 Apr 12;6(4):e94. doi: 10.2196/mhealth.9754. PMID 29650506
- [Background] Kubala AG, Barone Gibbs B, Buysse DJ, Patel SR, Hall MH, Kline CE. Field-based Measurement of Sleep: Agreement between Six Commercial Activity Monitors and a Validated Accelerometer. Behav Sleep Med. 2020 Sep-Oct;18(5):637-652. doi: 10.1080/15402002.2019.1651316. Epub 2019 Aug 27. PMID 31455144
- [Background] Gordt K, Gerhardy T, Najafi B, Schwenk M. Effects of Wearable Sensor-Based Balance and Gait Training on Balance, Gait, and Functional Performance in Healthy and Patient Populations: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Gerontology. 2018;64(1):74-89. doi: 10.1159/000481454. Epub 2017 Nov 1. PMID 29130977
- [Background] Kahawage P, Jumabhoy R, Hamill K, de Zambotti M, Drummond SPA. Validity, potential clinical utility, and comparison of consumer and research-grade activity trackers in Insomnia Disorder I: In-lab validation against polysomnography. J Sleep Res. 2020 Feb;29(1):e12931. doi: 10.1111/jsr.12931. Epub 2019 Oct 18. PMID 31626361
- [Background] de Zambotti M, Goldstone A, Claudatos S, Colrain IM, Baker FC. A validation study of Fitbit Charge 2 compared with polysomnography in adults. Chronobiol Int. 2018 Apr;35(4):465-476. doi: 10.1080/07420528.2017.1413578. Epub 2017 Dec 13. PMID 29235907
- [Background] Danzig R, Wang M, Shah A, Trotti LM. The wrist is not the brain: Estimation of sleep by clinical and consumer wearable actigraphy devices is impacted by multiple patient- and device-specific factors. J Sleep Res. 2020 Feb;29(1):e12926. doi: 10.1111/jsr.12926. Epub 2019 Oct 17. PMID 31621129
- [Background] Bravo P, Contreras A, Perestelo-Perez L, Perez-Ramos J, Malaga G. [Looking for a more participative healthcare: sharing medical decision making]. Rev Peru Med Exp Salud Publica. 2013 Oct-Dec;30(4):691-7. Spanish. PMID 24448951
- [Background] Peake JM, Kerr G, Sullivan JP. A Critical Review of Consumer Wearables, Mobile Applications, and Equipment for Providing Biofeedback, Monitoring Stress, and Sleep in Physically Active Populations. Front Physiol. 2018 Jun 28;9:743. doi: 10.3389/fphys.2018.00743. eCollection 2018. PMID 30002629
- [Background] Lee JM, Kim Y, Welk GJ. Validity of consumer-based physical activity monitors. Med Sci Sports Exerc. 2014 Sep;46(9):1840-8. doi: 10.1249/MSS.0000000000000287. PMID 24777201
- [Background] Bunce C. Correlation, agreement, and Bland-Altman analysis: statistical analysis of method comparison studies. Am J Ophthalmol. 2009 Jul;148(1):4-6. doi: 10.1016/j.ajo.2008.09.032. No abstract available. PMID 19540984
- [Background] de Zambotti M, Baker FC, Willoughby AR, Godino JG, Wing D, Patrick K, Colrain IM. Measures of sleep and cardiac functioning during sleep using a multi-sensory commercially-available wristband in adolescents. Physiol Behav. 2016 May 1;158:143-9. doi: 10.1016/j.physbeh.2016.03.006. Epub 2016 Mar 9. PMID 26969518
- [Background] Tilmanne J, Urbain J, Kothare MV, Wouwer AV, Kothare SV. Algorithms for sleep-wake identification using actigraphy: a comparative study and new results. J Sleep Res. 2009 Mar;18(1):85-98. doi: 10.1111/j.1365-2869.2008.00706.x. PMID 19250177
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Derived] Concheiro-Moscoso P, Groba B, Alvarez-Estevez D, Miranda-Duro MDC, Pousada T, Nieto-Riveiro L, Mejuto-Muino FJ, Pereira J. Quality of Sleep Data Validation From the Xiaomi Mi Band 5 Against Polysomnography: Comparison Study. J Med Internet Res. 2023 May 19;25:e42073. doi: 10.2196/42073. PMID 37204853
- [Derived] Concheiro-Moscoso P, Martinez-Martinez FJ, Miranda-Duro MDC, Pousada T, Nieto-Riveiro L, Groba B, Mejuto-Muino FJ, Pereira J. Study Protocol on the Validation of the Quality of Sleep Data from Xiaomi Domestic Wristbands. Int J Environ Res Public Health. 2021 Jan 27;18(3):1106. doi: 10.3390/ijerph18031106. PMID 33513712